CLINICAL TRIAL: NCT00454662
Title: Combination of OLMesartan and Calcium Channel Blocker or Low Dose Diuretics in High Risk Elderly Hypertensive Patients Study (COLM-Study)
Brief Title: Combination of OLMesartan and CCB or Low Dose Diuretics in High Risk Elderly Hypertensive Patients Study (COLM-Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: COLM Study Research Organization (Other)
Collaborators: Japan Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31-JAN-2007; COLM001
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension; Cardiovascular Disease; Diabetes
Keywords: Elderly; Hypertension; Cardiovascular Diseases; Angiotensin II Type 1 Receptor Blockers; Calcium Channel Blockers; Diuretics; Combination Drug Therapy; Diabetes
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Diabetes Mellitus | interventions — Olmesartan Medoxomil; Amlodipine; azelnidipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): olmesartan medoxomil, Calcium channel blockers (amlodipine, azelnidipine)
  Interventions: Drug: olmesartan medoxomil / amlodipine or azelnidipine
- 2 (Active Comparator): AT1 subtype angiotensin II receptor antagonist/low dose diuretic
  Interventions: Drug: olmesartan medoxomil / low dose thiazide type drug

INTERVENTIONS:
Drug: olmesartan medoxomil / amlodipine or azelnidipine — AT1 subtype angiotensin II receptor antagonist / calcium channel blocker : 5-40mg of olmesartan medoxomil / 2.5-5mg of amlodipine or 8-16mg of azelnidipine
  Arms: 1
Drug: olmesartan medoxomil / low dose thiazide type drug — AT1 subtype angiotensin II receptor antagonist / low dose diuretic : 5-40mg of olmesartan medoxomil / low dose thiazide type drug
  Arms: 2

SUMMARY:
The purpose of this study is to investigate which combination therapy is more effective in reducing the incidence of cardiovascular events in Japanese elderly high-risk hypertensive patients: AT1 subtype angiotensin II receptor antagonist/calcium channel blocker or AT1 subtype angiotensin II receptor antagonist/low dose diuretic.

DETAILED DESCRIPTION:
Recently, antihypertensive combination therapies have been recommended by various guidelines because of their additive effects. Combination therapies of AT1 subtype angiotensin II receptor antagonist and calcium channel blocker or low dose diuretic have shown pharmacological benefit. However, reduction of cardiovascular events and safety profile of these combination therapies under same level of antihypertensive target have not been investigated yet.

In this study, primary objective is to compare two combination therapies when antihypertensive target is 140/90mmHg in elderly hypertensive patients with high cardiovascular risk.

Further study details as provided by COLM-Study data center

Primary Outcomes: A composite of fatal and non-fatal cardiovascular events: Sudden death (death of endogenous origin within 24 hours after acute onset); Cerebrovascular events (new occurrence or recurrence of a cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage or transient ischemic attack); Coronary events (new occurrence or recurrence of a myocardial infarction, coronary revascularization[PCI or CABG], hospitalization for angina pectoris, hospitalization for heart failure); Renal dysfunction (doubling of serum creatinine and creatinine ≥2.0 mg/dl, end stage renal disease) Secondary Outcomes: All deaths; Death from cardiovascular events; Effects on glucose metabolism(fasting plasma glucose, postprandial glucose, new onset of diabetes mellitus); Incidence of primary outcomes events; New occurrence of atrial fibrillation; Safety; Proportion of the subjects who withdrew from the allocated treatment

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 65 years or older, and less than 85 years (at the time of informed consent), regardless of sex
* Systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg in a sitting position on two consecutive measurements at clinic during use of 1 or more antihypertensive medications.
* Systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg in a sitting position on two consecutive measurements at clinic without antihypertensive medication.
* Require at least one of the following medical history or risk factors
* Medical history

  * Cerebrovascular accident: cerebral infarction, brain hemorrhage, subarachnoid hemorrhage（6 months or more prior to registration）
  * Myocardial infarction, coronary revascularization (PCI or CABG) （6 months or more prior to registration）
  * Angina pectoris (except for the patients having history of hospitalization within 6 months prior to registration)
* Risk factors

  * Male
  * Current diabetes mellitus, fasting glucose ≥ 110mg/dL or postprandial glucose ≥ 140mg/dl
  * Hypercholesterolemia (Total cholesterol ≥ 260mg/dL)
  * Low HDL cholesterolemia (HDL-C <40mg/dL)
  * Microalbuminuria (albumin/cr ≥ 30mg/gCr) or proteinuria (protein ≥ 1＋)
  * Left ventricular hypertrophy (ST-T change in the ECG and SV1＋RV5 ≥ 35mm, or left ventricular mass index: male ≥ 125 g/m2, female ≥ 110 g/m2)

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* History of cerebrovascular accident (including TIA) or myocardial infarction within 6 months before registration
* Percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) done within 6 months before registration or scheduled
* History of hospitalization for angina pectoris or heart failure within 6 months before registration
* Severe heart failure (New York Heart Association [NYHA] functional class III or more severe)
* Complications of atrial fibrillation, atrial flutter or severe arrhythmia
* Severe hepatic or renal dysfunction (including current treatment of dialysis or renal dysfunction with serum creatinine ≥ 2.0mg/dL)
* Not appropriate for change to the study drugs from current therapy for concurrent disease including coronary diseases (i.e. calcium channel blockers, diuretics, etc)
* History of serious side effect from study drugs (AT1 subtype angiotensin II receptor antagonist, calcium channel blocker, diuretic)
* Life threatening condition (malignant tumor, etc)
* Not suited to be study subject judged by a study physician

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5141 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Composite of following events: Sudden death, Cerebrovascular events, Coronary events, Renal dysfunction | 3 to 4.5 years (duration of planned treatment phase)

SECONDARY OUTCOMES:
All deaths, Death from cardiovascular events, Glucose metabolism, Incidence of primary outcomes events, New onset of atrial fibrillation, Safety, Withdrawal rate | 3 to 4.5 years (duration of planned treatment phase)

CONTACTS AND LOCATIONS:
Overall Officials: Toshio Ogihara, MD, Study Chair — Emeritus Professor Osaka University; Takao Saruta, MD, Study Chair — Emeritus Professor Keio University
Locations (1):
- COLM-Study Data Center, Kamiyacho Mount Bld.14F, 4-3-20 Toranomon Minato-ku, Tokyo, Japan

REFERENCES:
- [Derived] Rakugi H, Ogihara T, Saruta T, Kawai T, Saito I, Teramukai S, Shimada K, Katayama S, Higaki J, Odawara M, Tanahashi N, Kimura G; COLM Investigators. Preferable effects of olmesartan/calcium channel blocker to olmesartan/diuretic on blood pressure variability in very elderly hypertension: COLM study subanalysis. J Hypertens. 2015 Oct;33(10):2165-72. doi: 10.1097/HJH.0000000000000668. PMID 26066644